CLINICAL TRIAL: NCT05300906
Title: The Effectiveness of Engagement-based Personalization of a Two-week Digital Mental Health Intervention Targeting Wellbeing: a Randomized Controlled Trial
Brief Title: The Effectiveness of Engagement-based Personalization of a Digital Mental Health Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Twente (Other)
Responsible Party: Principal Investigator, Saskia Kelders, Associate Professor, University of Twente
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Personalization Trial
Record Dates: First submitted 2022-03-03; First posted 2022-03-29 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Well-being

STUDY DESIGN:
Intervention Model Description: participants are randomized to either the personalized or the non-personalized intervention.
Masking Description: Participants will not be informed about their randomized condition (personalized or non-personalized), but it is likely that they will infer it from the intervention that they receive.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized (Experimental): Participants in the personalized arm will receive the optimal combination of content, feedback and design, based on their baseline engagement scores.
  Interventions: Behavioral: personalized 2-week mobile wellbeing intervention
- non-personalized (Active Comparator): Participants in the non-personalized arm will receive a randomly selected version of the 27 possible interventions, regardless of their baseline engagement scores.
  Interventions: Behavioral: non-personalized 2-week mobile wellbeing intervention

INTERVENTIONS:
Behavioral: personalized 2-week mobile wellbeing intervention — For the study, 27 versions of a 2-week mobile wellbeing intervention are created. These versions vary on content (Cognitive Behavioral Therapy, meaning, positive psychology), feedback (text, text with avatar, pre-recorded video) and design (non-gamified, competitively gamified, storyline gamified). At baseline, participants preview all variations and indicate their expected engagement. Participants in the personalized condition will receive the optimal combination of content, feedback and design, based on their baseline engagement scores.
  Each version of the intervention consists of a module per day. Each module contains psychoeducation and exercises based on content of the version. Moreover, each module contains pre-specified general feedback and supportive messages.
  Arms: Personalized
Behavioral: non-personalized 2-week mobile wellbeing intervention — For the study, 27 versions of a 2-week mobile wellbeing intervention are created. These versions vary on content (Cognitive Behavioral Therapy, meaning, positive psychology), feedback (text, text with avatar, pre-recorded video) and design (non-gamified, competitively gamified, storyline gamified). At baseline, participants preview all variations and indicate their expected engagement. Participants in the non-personalized condition will receive a random version of the intervention.
  Each version of the intervention consists of a module per day. Each module contains psychoeducation and exercises based on content of the version. Moreover, each module contains pre-specified general feedback and supportive messages.
  Arms: non-personalized

SUMMARY:
This study will investigate the effectiveness of an engagement-based personalized 2-week mobile wellbeing intervention, vs the effectiveness of a non-personalized 2-week mobile wellbeing intervention.

ELIGIBILITY:
Inclusion Criteria:

* at least mild depressive or anxiety complaints; >4 Generalized Anxiety Disorder 7-item scale OR Patient Health Questionnaire 9-item scale
* access to smartphone with internet
* adequate English literacy

Exclusion Criteria:

* none

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in wellbeing, measured with the Mental Health Continuum Short Form, at 3 weeks. | baseline, 3 weeks
  Wellbeing will be measured in an online survey, using the Mental Health Continuum Short Form. This validated scale consists of 14 items. The scale's total scores range from 14 to 84, with higher scores indicating higher wellbeing and thus better outcomes.
Change from baseline in depressive symptoms, measured with the Patient Health Questionnaire-9, at 3 weeks. | baseline, 3 weeks
  Depressive symptoms will be measured in an online survey, using the Patient Health Questionnaire-9. This validated scale consists of 9 items. The scale's total scores range from 0 to 27, with higher scores indicating higher depressive symptoms and thus worse outcomes.
Change from baseline in anxiety symptoms, measured with the Generalized Anxiety Disorder 7-item scale, at 3 weeks. | baseline, 3 weeks
  Depressive symptoms will be measured in an online survey, using the Generalized Anxiety Disorder 7-item scale. This validated scale consists of 6 items. The scale's total scores range from 0 to 21, with higher scores indicating higher anxiety symptoms and thus worse outcomes.

SECONDARY OUTCOMES:
Adherence | after 3 weeks
  Number of modules completed
Engagement, measured with the TWente Engagement with Ehealth Technologies Scale. | after 1 day
  Engagement will be measured within the intervention, with the validated TWente Engagement with Ehealth Technologies Scale. This is a 9 item scale, with a total score ranging from 0 to 36, with higher scores indicating higher engagement and thus better outcomes.
Engagement, measured with the TWente Engagement with Ehealth Technologies Scale. | after 7 days
  Engagement will be measured within the intervention, with the validated TWente Engagement with Ehealth Technologies Scale. This is a 9 item scale, with a total score ranging from 0 to 36, with higher scores indicating higher engagement and thus better outcomes.
Engagement, measured with the TWente Engagement with Ehealth Technologies Scale. | after 3 weeks
  Engagement will be measured within the intervention, with the validated TWente Engagement with Ehealth Technologies Scale. This is a 9 item scale, with a total score ranging from 0 to 36, with higher scores indicating higher engagement and thus better outcomes.
Change from baseline in wellbeing, measured with the Mental Health Continuum Short Form, at 8 weeks. | baseline, 8 weeks
  Wellbeing will be measured in an online survey, using the Mental Health Continuum Short Form. This validated scale consists of 14 items. The scale's total scores range from 14 to 84, with higher scores indicating higher wellbeing and thus better outcomes.
Change from baseline in depressive symptoms, measured with the Patient Health Questionnaire-9, at 8 weeks. | baseline, 8 weeks
  Depressive symptoms will be measured in an online survey, using the Patient Health Questionnaire-9. This validated scale consists of 9 items. The scale's total scores range from 0 to 27, with higher scores indicating higher depressive symptoms and thus worse outcomes.
Change from baseline in anxiety symptoms, measured with the Generalized Anxiety Disorder 7-item scale, at 8 weeks. | baseline, 8 weeks
  Depressive symptoms will be measured in an online survey, using the Generalized Anxiety Disorder 7-item scale. This validated scale consists of 6 items. The scale's total scores range from 0 to 21, with higher scores indicating higher anxiety symptoms and thus worse outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Saskia M Kelders, PhD, Principal Investigator — University of Twente
Locations (1):
- University of Twente, Enschede, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
The plan is to share anonymized data from the study in a open science database. Specifics are not yet established.